CLINICAL TRIAL: NCT04704050
Title: Effect of Dronedarone on Atrial Fibrosis Progression and Atrial Fibrillation Recurrence Post Ablation: The EDORA Trial
Brief Title: Effect of Dronedarone on Atrial Fibrosis Progression and Atrial Fibrillation Recurrence
Acronym: EDORA
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Sponsor withdrew funding
Sponsor: Tulane University School of Medicine (Other)
Collaborators: University of Washington (Other); Marrek, INC (Unknown); Sanofi (Industry); Preventice (Industry); Mckesson (Unknown)
Responsible Party: Sponsor
Organization: Tulane University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2830294
Record Dates: First submitted 2021-01-05; First posted 2021-01-11 (Actual); Results first posted 2025-10-16 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Atrial Fibrillation; Atrial Fibrillation Recurrent
Keywords: Atrial Fibrillation; Atrial Fibrillation Recurrent; Heart Murmur; Dronedarone; Atrial Fibrosis; Atrial Fibrosis Progression; Atrial Fibrosis Regression; Atrial Arrhythmia; Cardiac Arrhythmia; Cardiovascular Events; Multaq
MeSH Terms: conditions — Atrial Fibrillation; Heart Murmurs; Arrhythmias, Cardiac | interventions — Dronedarone; Tablets

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Treatment Group (Active Comparator): Dronedarone 400 mg orally, twice per day (BID)
  Interventions: Drug: dronedarone 400 mg Oral Tablet
- Control Group (Placebo Comparator): Placebo tablet orally, twice per day (BID)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: dronedarone 400 mg Oral Tablet — Dronedarone is an anti-arrhythmic drug with properties belonging to Vaughan-Williams class I-IV.
  Participants will receive dronedarone 400 mg tablet, to be taken orally and twice daily for 52 weeks.
  Other Names: Multaq®
  Arms: Treatment Group
Drug: Placebo — Participants will receive a placebo tablet matching the physical appearance of dronedarone, to be taken orally and twice daily for 52 weeks.
  Arms: Control Group

SUMMARY:
Patients who have undergone cardiac ablation will be randomized and blinded to one of two groups; one group will receive dronedarone while the other group will receive a placebo. The incidence of atrial fibrillation recurrence, as well as atrial fibrosis progression, will be analyzed between the two trial groups.

DETAILED DESCRIPTION:
The purpose of this trial is to determine whether dronedarone is effective in slowing the progression of fibrosis and decreasing atrial fibrillation recurrence in patients who have undergone ablation therapy.

Patients with atrial fibrillation (AF) undergoing ablation will be stratified by age and gender (>65 years and <65 years, male and female) as well as by type of atrial fibrillation (paroxysmal, persistent, etc.) and then randomized to one of two trial groups. They will either receive dronedarone 400 mg BID (twice daily) (treatment group) or placebo (control group). The control group will be started on placebo, and treating physicians will be advised to limit the initiation of anti-arrhythmic drugs (standard of care, SOC) to necessary cases only, avoiding amiodarone and dronedarone.

Each patient will receive a pre-ablation Cardiac Magnetic Resonance imaging (CMR) (SOC) scan, followed by scans at 3 and 12-month post-ablation. Quality of Life (QoL) changes will be evaluated from baseline and at 3 months and 12-months via the Atrial Fibrillation Effect on Quality-Of-Life (AFEQT) online questionnaire form. AF burden (frequency, duration and severity of an AF episode) if present, will be evaluated from baseline and at 3 months and 12-months via the Atrial Fibrillation Severity Scale (AFSS) online questionnaire form.

Patients will be followed post-ablation for AF recurrence and burden assessment with a continuous 30-day ECG wearable patch starting at discharge (SOC), then at 3,6,9 and 12 months post-ablation

Phone call visits will occur at 6 and 9 months to monitor for medication compliance as well as to assess that devices are working accordingly. Evaluation of adverse events (AE's) as well as whether a patient has reached any trial endpoints will be analyzed at this time.

Physicians will be advised to avoid adjustments in drug therapy unless necessary (severely symptomatic patients, patients with heart failure). Severely symptomatic patients will be defined as, patients with non-tolerated palpitations or chest pain, dizziness, syncope, dyspnea, or suddenly reduced ability to exercise.

Any initiation or change of an anti-arrhythmic treatment in the treatment or control group will be considered as a secondary endpoint. Patients will continue to be monitored for fibrosis progression and AF burden via CMR scans and ECG wearable devices until the end of the follow-up period. In the case of AF recurrence after ablation, anti-arrhythmic drugs (AAD) initiation or change will be left to the discretion of the treating physician.

ELIGIBILITY:
Inclusion Criteria: Patients must meet the following criteria to be enrolled in the trial.

* Male or female patients aged over 18 years of age.
* Patients with paroxysmal or persistent atrial fibrillation who are undergoing ablation of atrial fibrillation, regardless of whether they were receiving an anti-arrhythmic drug (AADs) before enrollment or not.

Exclusion Criteria: Patients will be excluded from enrollment if any of the following criteria are present.

* Any health-related gadolinium/MRI contraindications (e.g. allergy to gadolinium, pacemakers, Implantable Cardioverter Defibrillators [ICD's], other devices/implants contraindicated for use of MRI, etc.).
* Patients weighing >300 Ibs. (MRI quality decreases as BMI increases).
* Patients with contraindications to dronedarone. (Including patients with decompensated heart failure or class NYHA IV (New York Heart Association Class IV), second or third-degree atrioventricular (AV) block or sick-sinus syndrome [except when used in conjunction with a functioning pacemaker]), concomitant use of strong cytochrome P450, family 3, subfamily A (CYP-3A) inhibitors or other Class I or III AADs, drug or herbal products that prolongs the QT interval and may induce Torsades de Pointes.
* Liver or lung toxicity related to the previous use of amiodarone, severe hepatic impairment including any stage of cirrhosis and acute liver failure, bradycardia <50bpm, QTc Bazett interval >500ms or PR interval >280ms, or hypersensitivity to the active substance or to any of its excipients.
* Acute or chronic severe renal disease with a low glomerular filtration rate (GFR), <30 mL per minute per 1.73m2 will be excluded from the trial.
* Patients with a history of prior left atrial ablation or valvular cardiac surgery (myocardial scarring/fibrosis from prior surgeries may confound data).
* Pre-menopausal (last menstruation <1 year prior to screening) who:

  1. are pregnant or breast-feeding or plan to become pregnant during the study period or,
  2. are not surgically sterile or,
  3. are of childbearing potential and not practising two acceptable methods of birth control or,
  4. do not plan to continue practising two acceptable methods of birth control throughout the trial (highly effective methods of birth control are defined as those, used alone, or in combination, that result in a low failure rate i.e. less than 1% per year when used consistently and correctly).
* Patients who do not have access to the Internet/e-mail.
* Patients without daily access to a smart phone-compatible with ECG Check device application and ability to upload ECG tracings for the entire follow-up period.
* Patients unable or unwilling to return to the clinic for follow up CMR scans.
* Patients with cognitive impairments who are unable to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Participant eligibility is based on the self-representation of gender identity.
Enrollment: 22 (Actual)
Dates: Start 2021-05-15 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2022-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nassir F Marrouche, MD, Principal Investigator — Tulane University School of Medicine
Locations (4):
- United States (4):
  - University of Colorado Health Memorial, Colorado Springs, Colorado
  - Emory University, Atlanta, Georgia
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hagens VE, Ranchor AV, Van Sonderen E, Bosker HA, Kamp O, Tijssen JG, Kingma JH, Crijns HJ, Van Gelder IC; RACE Study Group. Effect of rate or rhythm control on quality of life in persistent atrial fibrillation. Results from the Rate Control Versus Electrical Cardioversion (RACE) Study. J Am Coll Cardiol. 2004 Jan 21;43(2):241-7. doi: 10.1016/j.jacc.2003.08.037. PMID 14736444
- [Background] Blomstrom-Lundqvist C, Gizurarson S, Schwieler J, Jensen SM, Bergfeldt L, Kenneback G, Rubulis A, Malmborg H, Raatikainen P, Lonnerholm S, Hoglund N, Mortsell D. Effect of Catheter Ablation vs Antiarrhythmic Medication on Quality of Life in Patients With Atrial Fibrillation: The CAPTAF Randomized Clinical Trial. JAMA. 2019 Mar 19;321(11):1059-1068. doi: 10.1001/jama.2019.0335. PMID 30874754
- [Background] Marrouche NF, Brachmann J, Andresen D, Siebels J, Boersma L, Jordaens L, Merkely B, Pokushalov E, Sanders P, Proff J, Schunkert H, Christ H, Vogt J, Bansch D; CASTLE-AF Investigators. Catheter Ablation for Atrial Fibrillation with Heart Failure. N Engl J Med. 2018 Feb 1;378(5):417-427. doi: 10.1056/NEJMoa1707855. PMID 29385358
- [Background] Packer DL, Mark DB, Robb RA, Monahan KH, Bahnson TD, Poole JE, Noseworthy PA, Rosenberg YD, Jeffries N, Mitchell LB, Flaker GC, Pokushalov E, Romanov A, Bunch TJ, Noelker G, Ardashev A, Revishvili A, Wilber DJ, Cappato R, Kuck KH, Hindricks G, Davies DW, Kowey PR, Naccarelli GV, Reiffel JA, Piccini JP, Silverstein AP, Al-Khalidi HR, Lee KL; CABANA Investigators. Effect of Catheter Ablation vs Antiarrhythmic Drug Therapy on Mortality, Stroke, Bleeding, and Cardiac Arrest Among Patients With Atrial Fibrillation: The CABANA Randomized Clinical Trial. JAMA. 2019 Apr 2;321(13):1261-1274. doi: 10.1001/jama.2019.0693. PMID 30874766
- [Background] Marrouche NF, Wilber D, Hindricks G, Jais P, Akoum N, Marchlinski F, Kholmovski E, Burgon N, Hu N, Mont L, Deneke T, Duytschaever M, Neumann T, Mansour M, Mahnkopf C, Herweg B, Daoud E, Wissner E, Bansmann P, Brachmann J. Association of atrial tissue fibrosis identified by delayed enhancement MRI and atrial fibrillation catheter ablation: the DECAAF study. JAMA. 2014 Feb 5;311(5):498-506. doi: 10.1001/jama.2014.3. PMID 24496537
- [Background] Kheirkhahan M, Baher A, Goldooz M, Kholmovski EG, Morris AK, Csecs I, Chelu MG, Wilson BD, Marrouche NF. Left atrial fibrosis progression detected by LGE-MRI after ablation of atrial fibrillation. Pacing Clin Electrophysiol. 2020 Apr;43(4):402-411. doi: 10.1111/pace.13866. PMID 31867751
- [Background] Hohnloser SH, Crijns HJ, van Eickels M, Gaudin C, Page RL, Torp-Pedersen C, Connolly SJ; ATHENA Investigators. Effect of dronedarone on cardiovascular events in atrial fibrillation. N Engl J Med. 2009 Feb 12;360(7):668-78. doi: 10.1056/NEJMoa0803778. PMID 19213680
- [Background] Akoum N, Fernandez G, Wilson B, Mcgann C, Kholmovski E, Marrouche N. Association of atrial fibrosis quantified using LGE-MRI with atrial appendage thrombus and spontaneous contrast on transesophageal echocardiography in patients with atrial fibrillation. J Cardiovasc Electrophysiol. 2013 Oct;24(10):1104-9. doi: 10.1111/jce.12199. Epub 2013 Jul 11. PMID 23844972
- [Derived] Marrouche NF, Dagher L, Wazni O, Akoum N, Mansour M, El Hajjar AH, Bhatnagar A, Hua H; EDORA Investigators. Effect of DrOnedarone on atrial fibrosis progression and atrial fibrillation recurrence postablation: Design of the EDORA randomized clinical trial. J Cardiovasc Electrophysiol. 2021 Dec;32(12):3203-3210. doi: 10.1111/jce.15274. Epub 2021 Nov 2. PMID 34664772

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Group: Dronedarone 400 mg orally, twice per day (BID)
  dronedarone 400 mg Oral Tablet: Dronedarone is an anti-arrhythmic drug with properties belonging to Vaughan-Williams class I-IV.
  Participants will receive dronedarone 400 mg tablet, to be taken orally and twice daily for 52 weeks.
Period: Overall Study
Arm/Group | Treatment Group | Control Group
Started | 12 | 10
Completed | 6 | 7
Not Completed | 6 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Group | Control Group | Total
Number analyzed (Participants) | 12 | 10 | 22
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 66 [55.25 to 78.25] | 64.50 [52.50 to 69.75] | 66 [53.75 to 72.50]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 6 | 5 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 10 | 9 | 19
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 12 | 10 | 22

OUTCOME MEASURES:

1. Primary Outcome: Post-ablation Atrial Fibrillation Recurrence
Description: Investigators monitored subjects upon discharge, 24-48 hours after AF ablation. This was recorded by either the occurrence of a single positive atrial arrhythmias (AA) ECG reading on a 12-lead ECG, Holter monitor, obtained on the daily event strips from the Preventice monitoring device, or 30-day monitoring patch.
Time Frame: Up to 56 weeks. From date of ablation until the date of first documented Atrial Fibrillation recurrence, whichever came first, assessed up to 56 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 12 | 10
Participants | 2 | 1

2. Primary Outcome: Post-ablation Atrial Fibrillation Recurrence Documented by an AAD Initiation
Description: New anti-arrhythmic drug (AAD) initiation for AF recurrence after AF ablation, including initiation of the treatment during the blanking period, or with no available positive ECG reading.
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 12 | 10
Participants | 1 | 2

3. Secondary Outcome: Atrial Fibrillation Episodes
Description: Atrial arrhythmia (AA) episodes associated with palpitations, chest pain, dyspnea, dizziness, syncope, or unusual fatigue and weakness were assessed using the Atrial Fibrillation Severity Scale (AFSS) questionnaire. The AFSS is a validated questionnaire designed to measure the burden of atrial arrhythmias, including atrial fibrillation and other irregular heart rhythms. The AA symptom burden score is derived from the AFSS summary score, which averages the frequency, duration, and patient-perceived severity of AA episodes.
  The AFSS symptom burden score ranges from 3 to 30, with higher scores indicating greater AA burden. Subscale scores (frequency, duration, and severity) are each rated on a scale of 1 to 10 and are averaged to calculate the total burden score.
  Patients completed the AFSS at baseline, 3 months, and 12 months. Reported data in the results table reflect the mean score at the 12-month time point.
Time Frame: At baseline, at month 3, at month 12
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 12 | 10
Scores on a scale | 7.5 (1.73) | 7.8 (2.17)

4. Secondary Outcome: Repeat Cardiac Ablation
Description: Whether patients in either treatment arm require a repeat cardiac ablation.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 12 | 10
Participants | 1 | 0

5. Secondary Outcome: Cardioversion
Description: Whether patients in either treatment arm require cardioversion.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 12 | 10
Participants | 2 | 1

6. Secondary Outcome: Atrial Fibrillation Burden
Description: The percentage of time a patient is in atrial fibrillation during the monitoring period, 24-48 hours and, at 3 months and 12 months post-ablation. Burden will be recorded as a time-weighted average (%) based on data from wearable devices.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: Percentage of time
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 12 | 10
Percentage of time | 9 (4.55) | 4.5 (5.8)

7. Secondary Outcome: Quality of Life (Online Questionnaire Form)
Description: Quality of life (QoL) was assessed through the Atrial Fibrillation Severity Scale (AFSS), a validated instrument that evaluates the impact of AF across multiple domains, including symptom burden, health care utilization, and overall well-being.
  The Global Well-being domain of the AFSS is assessed using a single-item question (A4), which measures overall quality of life on a scale from 1 to 10, where higher scores indicate better quality of life.
  Patients completed the questionnaire at baseline, 3 months, and 12 months. The reported data in the results table reflect the mean score at the 12-month time point.
Time Frame: At baseline, at month 3, at month 12
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 12 | 10
Scores on a scale | 8.8 (1.30) | 10 (0)

8. Secondary Outcome: Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]
Description: Assessment of adverse events related to treatment given. Evaluated at 3, 12 months visits and during 6 & 9 month phone call visits.
Time Frame: Through trial completion, up to 56 weeks.
Measure: Number; unit: Events
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 12 | 10
Events
  Anemia | 1 | 0
  Fatigue | 1 | 0
  Hypoxemia | 1 | 0
  Elevated creatinine | 1 | 0
  Thrombocytopenia | 1 | 0
  Dyspnea | 1 | 0
  Dyspnea on effort | 1 | 0
  Increased Troponin | 1 | 0
  Intermittent Nausea | 1 | 0
  Intermittent Headache | 1 | 0
  Upset Stomach | 1 | 0
  Right shoulder pain | 1 | 0
  Right rotator cuff tear | 1 | 0
  Elevated uric acid levels | 0 | 1
  Excessive flatulence | 0 | 1
  Hemorrhoids | 1 | 0
  Prostate hyperplasia | 1 | 0
  Hypertension | 0 | 1
  Worsening of Hyperlipidemia | 0 | 1
  Right lung mass | 0 | 1
  Increased shoulder pain | 0 | 1
  Leukocytosis | 0 | 1
  Nausea | 1 | 0
  Diarrhea | 1 | 0
  Rash on Chest | 1 | 0
  Spinal Stenosis | 1 | 0
  Urinary incontinence | 1 | 0
  Erectile dysfunction | 1 | 0

9. Other Pre Specified Outcome: Hospitalization
Description: Records of any cardiac events requiring hospitalization.
Time Frame: 1 year
Measure: Number; unit: Events
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 12 | 10
Events
  Anemia | 1 | 0
  Chest Pain | 0 | 1
  Dizziness | 0 | 1
  Dyspnea | 0 | 1
  Hematuria | 0 | 1
  GERD | 0 | 1
  Peripheral neuropathy | 1 | 0
  Increased Troponin | 1 | 0
  Right lower extremity swelling | 0 | 1
  Left lower extremity swelling | 0 | 1
  Left upper extremity swelling | 0 | 1
  Acute gout flare-up | 0 | 1
  Cellulitis | 0 | 1
  Fluid Overload | 0 | 1
  Acute Kidney Injury | 0 | 1
  Acute Tubular Necrosis | 0 | 1
  Hyperkalemia | 0 | 1
  Hypotension | 0 | 1

10. Other Pre Specified Outcome: Mortality
Description: Records of mortality associated with cardiovascular events.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 12 | 10
Participants | 0 | 0

11. Other Pre Specified Outcome: Stroke/ Transient Ischemic Attacks (TIA)
Description: Records of stroke or TIA based on cardiac emboli.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 12 | 10
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 13 Months
Arm/Group | Treatment Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/10
Serious Adverse Events (participants affected / at risk) | 2/12 | 3/10
Other Adverse Events (participants affected / at risk) | 2/12 | 3/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group (N=12) | Control Group (N=10)
Hospitalization (Cardiac disorders) | 2 (3) | 3 (15) — Hospitalization
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Dizziness (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Dyspnea (Cardiac disorders) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
GERD (Gastrointestinal disorders) | 0 (0) | 1 (1)
Peripheral neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Increased Troponin (Cardiac disorders) | 1 (1) | 0 (0)
Chest Pain (Cardiac disorders) | 0 (0) | 1 (1)
Right lower extremity swelling (Vascular disorders) | 0 (0) | 1 (1)
Left lower extremity swelling (Vascular disorders) | 0 (0) | 1 (1)
Left upper extremity swelling (Vascular disorders) | 0 (0) | 1 (1)
Acute gout flare-up (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cellulitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Fluid Overload (Cardiac disorders) | 0 (0) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Acute Tubular Necrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypotension (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group (N=12) | Control Group (N=10)
Hypertension (Cardiac disorders) | 0 (0) | 1 (1)
Worsening of Hyperlipidemia (Cardiac disorders) | 0 (0) | 1 (1)
Dyspnea (Cardiac disorders) | 1 (1) | 0 (0)
Dyspnea on effort (Cardiac disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Elevated Creatinine (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Prostate hyperplasia (Renal and urinary disorders) | 1 (1) | 0 (0)
Hypoxemia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Right lung mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Intermittent Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upset Stomach (Gastrointestinal disorders) | 1 (1) | 0 (0)
Excessive flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intermittent Headache (Nervous system disorders) | 1 (1) | 0 (0)
Fatigue (Nervous system disorders) | 1 (1) | 0 (0)
Right shoulder pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Right rotator cuff tear (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Increased shoulder pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Elevated uric acid levels (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rash on Chest (General disorders) | 1 (1) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Early termination and incomplete data collections for several outcome measures. All data that was collected was added to the results section for this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-27): https://cdn.clinicaltrials.gov/large-docs/50/NCT04704050/Prot_SAP_000.pdf